CLINICAL TRIAL: NCT04691609
Title: Assiut University Registry for ACS Patients During COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah ObiedAllah Fouad, Principal investigator, Assiut University
Other Study IDs: ACS in COVID-19 era
Record Dates: First submitted 2020-09-21; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: ACS-COVID-19-Assiut

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To register pathological events occurring to all acute coronary syndrome patients coming to Assiut university heart hospital through one year during COVID- 19 pandemic

DETAILED DESCRIPTION:
In the face of the quickly evolving coronavirus disease 2019 (COVID-19) pandemic, many health-care systems around the globe have modified their routine management of patients presenting with acute cardiovascular emergencies including patients with ACS.A unifying theme in the new management strategies is the adoption of new restrictive measures to meet the challenges of increased risk of infection of health-care workers; limited numbers of beds, shortage of personal protective equipment (PPE), inadequate number of protected catheterization rooms; and the clinical overlap between ACS and COVID-19 infection in some of patients.

In developing countries, with an already strained health system due to economic problems, the situation is more challenging and needs the formulation of efficient protocols that can accommodate several medical and socioeconomic challenges.

Egypt, with an estimated population of 100 million, is facing exceptional challenges during the COVID-19 crisis. Because large scale use of polymerase chain reaction (PCR) test for SARS-CoV-2 in a large population is a problem, the prevalence of COVID-19 infection in Egypt is unknown. Furthermore, the supply of PPE falls far short of demands with lack of professionally protected cardiac catheterization rooms. With progression of the pandemic in such a large population, care of COVID-19 patients is expected to rapidly overwhelm the supplies, beds, and staff available in Egyptian hospitals.

The Cardiology Department in Assiut university hospital has revised the management protocols for ACS patients and implemented new management protocols both for patients with ST-segment elevation myocardial infarction (STEMI) and Non-ST-segment elevation acute coronary syndromes (NSTE-ACS).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms or ECG indicative of acute coronary syndrome admitted to Assiut heart hospital

Exclusion Criteria:

* The only exclusion criteria is refusal of the patient to participate in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: ACS patients admitted to Assiut university heart hospital either male or female, young or old, COVID-19 confirmed, suspected or even excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Main Number, distribution and oucome of all ACS patients coming to Assiut heart hospital | about 1 year
  Number, distribution and outcome of all ACS patients coming to Assiut heart hospital(as age, gender, risk factors of coronary artery diseases and their effect on incidence and progress of ACS )

SECONDARY OUTCOMES:
To register pathological events occurring to all acute coronary syndrome patients coming to Assiut university heart hospital through one year during COVID- 19 pandemic | about 1 year
  To evaluate clinical symptoms and signs of COVID -19 and acute coronary syndrome(Type of ACS, type of intervention or treatment for each case,complications if peresent, COVID - 19 status and if it affects ACS patient or not and follow up after 3 months and 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Khairy Hassan, Lecturer, Study Director — aymankhairy11@gmail.com
Locations (1):
- Samah ObiedAllah Fouad, Asyut, Resident, Egypt